CLINICAL TRIAL: NCT06327854
Title: Study of the Relationship Between Dietary Aspects and Oral Hygiene in Patients Undergoing Orthopedic Surgery
Brief Title: NUtrition and ORal Health in Orthopaedic Surgery
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: NUOROS (PI: M Briguglio); L4175 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Orthopedic Disorder; Metabolism and Nutrition Disorder
MeSH Terms: conditions — Musculoskeletal Diseases; Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This prospective observational study evaluates the relationship between the objective oral health status and the patient reported diet in 64 adult patients undergoing elective major orthopaedic surgery (hip, knee, or spine surgery).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥55
* Male and female gender
* Major elective orthopedic surgery (hip, knee, spinal)
* Signature of the informed consent

Exclusion Criteria:

* Inability to follow the study protocol
* Neuropsychiatric disease, developmental disorders

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients undergoing elective major orthopedic surgery, such as hip, knee, or spine surgery.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Association between pre-operative oral health and diet | Day before surgery
  Relationship between the objective oral health and the patient reported dietary score evaluated at hospital admission before major orthopedic surgery

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Briguglio, Principal Investigator — I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio
Locations (1):
- I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided